CLINICAL TRIAL: NCT03096951
Title: Prehabilitation Before Surgery in Colorectal Cancer With Improved Fast Track Rehabilitation : Part 1
Brief Title: Prehabilitation in Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, G.Reychler, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Part 1
Record Dates: First submitted 2017-03-17; First posted 2017-03-30 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Preoperative Exercise; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation group (Experimental): Preoperative and postoperative telerehabilitation
  Interventions: Behavioral: Prehabilitation
- Rehabilitation group (Active Comparator): Postoperative telerehabilitation
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Behavioral: Prehabilitation — Prehabilitation group will receive a 4-week tele-supervised prehabilitation and a 8-week tele-supervised postoperative rehabilitation.
  Arms: Prehabilitation group
Other: Rehabilitation — Rehabilitation group will receive World Health Organization recommendations on physical activity for health before surgery and a 8-week tele-supervised postoperative rehabilitation.
  Arms: Rehabilitation group

SUMMARY:
Objectives To investigate the impact of tele-supervised prehabilitation on functional capacity in colon cancer patients undergoing colorectal resection for cancer and to evaluate the effects of prehabilitation on muscle strength and endurance, quality of life (QoL), executive functions, fatigue and inflammatory and metabolic parameters.

Methods A randomized controlled trial will be conducted. Patients will be randomised into either a prehabilitation group or a control group. The prehabilitation group will receive tele-supervised prehabilitation for 4weeks and telerehabilitation for 8weeks post-surgery while control group will begin telerehabilitation only after surgery for 8weeks. Patients will care with an enhanced recovery pathway. Telerehabilitation pre and post-surgery will consist of three moderate-intensity aerobic and resistance sessions per week. Subjects will be assessed at baseline, pre-intervention, post-intervention and post-rehabilitation. The primary outcome will be functional capacity measured using the 6-min walk test. The secondary outcomes will be: physical measurement, quality of life, level of physical activity, executive functions, fatigue, body composition, blood test, energy expenditure.

DETAILED DESCRIPTION:
Study objectives Primary objective: The investigators want to assess if a tele-supervised prehabilitation improves preoperative cardio-respiratory fitness in colon cancer patients in the setting of an enhanced recovery pathway.

Secondary objectives

* The investigators want to examine if this tele-supervised prehabilitation has beneficial effects on muscle strength and endurance, on quality of life, on executive functions, on fatigue, on inflammatory parameters and on metabolic disruption pre-surgery.
* The investigators want to determine whether changes in the preoperative period remain in the postoperative period after 8 weeks of telerehabilitation.

Rationale and scientific background:

In Belgium, colon cancer is the third most common cancer in men and the second most common in women and is the second cause of cancer death. Surgery is currently the primary treatment for stage I to III. This surgery benefits from several years of multimodal program, commonly called "Fast Track" program or enhanced recovery. Nowadays, the lack of preoperative fitness is not specifically taken into account in the Fast Track program. Nevertheless, studies have shown that patients with poor preoperative physical fitness are less able to cope with the adverse effects of surgery and hospitalization resulting in increased risk of mortality, postoperative complications and functional recovery time. It seems relevant to intervene during the preoperative period to improve the patient's functional capacity before the surgery, via physical training to overcome the stress of the surgery and to improve postoperative recovery. This process is called "prehabilitation" Structured and supervised programs have shown to be effective and feasible. However, time, resources, expensive care are often a barrier for the patient. Thereby, a home-based tele-supervising rehabilitation would be an attractive therapeutic option to offer a distinct advantage in this regard. More specifically, "telerehabilitation can be defined as the application of telecommunication, remote sensing and operation technologies, and computing technologies to assist with the provision of medical rehabilitation services at a distance".

Study design A single-blind, randomized, controlled trial will be conducted. Participants will be randomized into either a prehabilitation group or a rehabilitation group. Participants in both groups will care in an Fast Track Program. An assessor who will be blinded to group allocation will collect outcomes measures for each participant.

To be eligible for this study participants will need to meet the following criteria: Diagnosis of colon cancer requiring surgery; more than 50 years of age; autonomous and voluntary person; able to read, write and understand French; Participants will be excluded if the participants have a physical impairment that would seriously impair physical mobility; have an unfavorable familial context; have a stoma; have an American Society of Anesthesiologists score IV-V; the surgery is an emergency; have neuropsychiatric disease.

Participants allocated to the prehabilitation group will undertake a telerehabilitation program that will start 4 weeks before the surgery and will continue during 8 weeks after the surgery. Participants in the control group will receive World Health Organization recommendations on physical activity for health before surgery. After the surgery, The control group will undertake a telerehabilitation program over an 8-week period.

The telerehabilitation program will combine aerobic and resistance training three sessions per week. Each 60-min session will begin and end with a five-minute warm-up/cool. The warm-up will be followed by 25 minutes of aerobic training. Aerobic exercise can include brisk walking, jogging, cycling, or swimming according to patient's preference. The intensity of the exercise was set between 60 à 75% of maximum heart rate (maximal heart rate=220 - age). And between 12 and 16 on Borg's Rating of Perceived Exertion Scale. Each participant will wear a heart monitor. The aerobic training will be followed by resistance exercise performed on eight exercises targeting major muscle groups (abdominal, hamstring, quadriceps, triceps, gluteus maximus, paraspinal muscles and shoulder muscles). Intensity must be between 12 and 16 on the Borg's Rating of Perceived Exertion Scale. A physiotherapist will provide detailed information about the program. The patient will receive a brochure in which there will be descriptions and pictures of exercises and a video including the resistance program was recorded on a website. The researcher will conduct weekly telephone calls with the participants. The aim of these calls will be to solve any problems of carrying out the training sessions and to discuss about possible adverse events. Moreover, the researcher will give messages of support and encouragement to improve adherence to the program.

Outcome measures will be assessed at four time points: at baseline (T0), one day before the scheduled date of surgery (T1), one week after the intervention (T2) and at the end of the postoperative rehabilitation (T3).

Primary outcome will be cardiorespiratory fitness 6min walk test). Secondary outcomes will be muscle strength and endurance (isokinetic dynamometer and 1min sit-to-stand-test), quality of life ("Euroquol-5D-3L" questionnaire); level of physical activity (International Physical Activity Questionnaire Short Form); fatigue (Functional Assessment of Cancer Therapy: Fatigue); executive functions (Trail Making test, Stroop test and fluency) ; blood test (neutrophil lymphocyte ratio, C reactive protein, fasting glucose, fasting insulin and cholesterol will be measured by bioelectrical impedance analysis); energy expenditure ("Sensewear®" armband).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colon cancer requiring surgery;
* more than 40 years of age;
* autonomous and voluntary person;
* able to read, write and understand French;
* Frailty phenotype criteria < 3

Exclusion Criteria:

* a physical impairment that would seriously impair physical mobility;
* an unfavorable familial context;
* a stoma;
* American Society of Anesthesiologists score IV-V;
* emergency;
* neuropsychiatric disease.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change in cardiorespiratory fitness | Assessments at baseline, one day before the surgery, 1 week after the surgery and immediately after the rehabilitation
  Cardiorespiratory is measured by a 6-minute walk test

SECONDARY OUTCOMES:
Change in muscle strength | Assessments at baseline, one day before the surgery, immediately after the rehabilitation
  Muscle strength is measured by using an isokinetic dynamometer
Change in muscle endurance | Assessments at baseline, one day before the surgery, 1week after the surgery and immediately after the rehabilitation
  Muscle endurance is measured by using the "1-minute sit-to-stand-test" (number of sit-to-stand cycles during 1 minute)
Change in quality of life | Assessments at baseline, one day before the surgery, 1week after the surgery and immediately after the rehabilitation
  Quality of life is measured by using the Euroquol-5D-3L questionnaire
Change in fatigue | Assessments at baseline, one day before the surgery, 1week after the surgery and immediately after the rehabilitation
  Fatigue is measured by using the Functional Assessment of Cancer Therapy: Fatigue questionnaire
Change in level of physical activity | Assessments at baseline, one day before the surgery, 1week after the surgery and immediately after the rehabilitation
  Level of physical activity is measured by using the International Physical Activity Questionnaire Short Form
Change in executive functions | Assessments at baseline, one day before the surgery, 1 week after the surgery and immediately after the rehabilitation
  Executive functions is measured by using the Trail Making test
Change in executive functions | Assessments at baseline, one day before the surgery, 1 week after the surgery and immediately after the rehabilitation
  Executive functions is measured by using the Fluency test
Change in weight | Assessments at baseline, one day before the surgery, 1 week after the surgery and immediately after the rehabilitation
  Weight (kg) is measured by using a bioelectrical impedance analysis
Change in lean body mass | Assessments at baseline, one day before the surgery, 1 week after the surgery and immediately after the rehabilitation
  Lean body mass (kg) is measured by using a bioelectrical impedance analysis
Change in fat body mass | Assessments at baseline, one day before the surgery, 1 week after the surgery and immediately after the rehabilitation
  Fat body mass (kg) is measured by using a bioelectrical impedance analysis
Energy expenditure | During 7 days before the surgery and during 7 days after the surgery
  Sensewear Armband
Change in Fasting glucose | Assessments at baseline, one day before the surgery, 1 week after the surgery and immediately after the rehabilitation
  Fasting glucose is measured by a blood test
Change in Fasting insulin | Assessments at baseline, one day before the surgery, 1 week after the surgery and immediately after the rehabilitation
  Fasting insulin is measured by a blood test
Change in cholesterol | Assessments at baseline, one day before the surgery, 1 week after the surgery and immediately after the rehabilitation
  Cholesterol is measured by a blood test
Change in neutrophil/lymphocyte | Assessments at baseline, one day before the surgery, 1 week after the surgery and immediately after the rehabilitation
  Neutrophil/lymphocyte is measured by a blood test
Change in C-reactive protein | Assessments at baseline, one day before the surgery, 1 week after the surgery and immediately after the rehabilitation
  C-reactive protein is measured by a blood test
Adherence | Assessments at baseline, one day before the surgery, 1 week after the surgery and immediately after the rehabilitation
  Percentage of sessions completed

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Woluwé-Saint-Lambert, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferlay J, Steliarova-Foucher E, Lortet-Tieulent J, Rosso S, Coebergh JW, Comber H, Forman D, Bray F. Cancer incidence and mortality patterns in Europe: estimates for 40 countries in 2012. Eur J Cancer. 2013 Apr;49(6):1374-403. doi: 10.1016/j.ejca.2012.12.027. Epub 2013 Feb 26. PMID 23485231
- [Background] Boereboom C, Doleman B, Lund JN, Williams JP. Systematic review of pre-operative exercise in colorectal cancer patients. Tech Coloproctol. 2016 Feb;20(2):81-9. doi: 10.1007/s10151-015-1407-1. Epub 2015 Nov 27. PMID 26614304
- [Background] Pallis AG, Papamichael D, Audisio R, Peeters M, Folprecht G, Lacombe D, Van Cutsem E. EORTC Elderly Task Force experts' opinion for the treatment of colon cancer in older patients. Cancer Treat Rev. 2010 Feb;36(1):83-90. doi: 10.1016/j.ctrv.2009.10.008. Epub 2009 Nov 26. PMID 19944536
- [Background] Nicholson A, Lowe MC, Parker J, Lewis SR, Alderson P, Smith AF. Systematic review and meta-analysis of enhanced recovery programmes in surgical patients. Br J Surg. 2014 Feb;101(3):172-88. doi: 10.1002/bjs.9394. PMID 24469618
- [Background] Fearon KC, Ljungqvist O, Von Meyenfeldt M, Revhaug A, Dejong CH, Lassen K, Nygren J, Hausel J, Soop M, Andersen J, Kehlet H. Enhanced recovery after surgery: a consensus review of clinical care for patients undergoing colonic resection. Clin Nutr. 2005 Jun;24(3):466-77. doi: 10.1016/j.clnu.2005.02.002. Epub 2005 Apr 21. PMID 15896435
- [Background] Wilson RJ, Davies S, Yates D, Redman J, Stone M. Impaired functional capacity is associated with all-cause mortality after major elective intra-abdominal surgery. Br J Anaesth. 2010 Sep;105(3):297-303. doi: 10.1093/bja/aeq128. Epub 2010 Jun 23. PMID 20573634
- [Background] Robinson TN, Wu DS, Pointer L, Dunn CL, Cleveland JC Jr, Moss M. Simple frailty score predicts postoperative complications across surgical specialties. Am J Surg. 2013 Oct;206(4):544-50. doi: 10.1016/j.amjsurg.2013.03.012. Epub 2013 Jul 20. PMID 23880071
- [Background] Lawrence VA, Hazuda HP, Cornell JE, Pederson T, Bradshaw PT, Mulrow CD, Page CP. Functional independence after major abdominal surgery in the elderly. J Am Coll Surg. 2004 Nov;199(5):762-72. doi: 10.1016/j.jamcollsurg.2004.05.280. PMID 15501119
- [Background] West MA, Lythgoe D, Barben CP, Noble L, Kemp GJ, Jack S, Grocott MP. Cardiopulmonary exercise variables are associated with postoperative morbidity after major colonic surgery: a prospective blinded observational study. Br J Anaesth. 2014 Apr;112(4):665-71. doi: 10.1093/bja/aet408. Epub 2013 Dec 8. PMID 24322573
- [Background] Debes C, Aissou M, Beaussier M. [Prehabilitation. Preparing patients for surgery to improve functional recovery and reduce postoperative morbidity]. Ann Fr Anesth Reanim. 2014 Jan;33(1):33-40. doi: 10.1016/j.annfar.2013.12.012. Epub 2014 Jan 17. French. PMID 24440732
- [Background] Spanjersberg WR, Reurings J, Keus F, van Laarhoven CJ. Fast track surgery versus conventional recovery strategies for colorectal surgery. Cochrane Database Syst Rev. 2011 Feb 16;(2):CD007635. doi: 10.1002/14651858.CD007635.pub2. PMID 21328298
- [Background] Cooper RA, Fitzgerald SG, Boninger ML, Brienza DM, Shapcott N, Cooper R, et al. Telerehabilitation: Expanding access to rehabilitation expertise. Proceedings of the IEEE. 2001;89(8):1174-93.
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub3. PMID 37162250
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2022 May 19;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub2. PMID 35588252